CLINICAL TRIAL: NCT07306637
Title: Wenjuanxing-Based Multidimensional Etiologic Screening and Clinical Validation of Chronic Cough in Children
Status: Not yet recruiting | Type: Observational
Sponsor: Shanghai Children's Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: SCMCIRB-YJ2025012
Record Dates: First submitted 2025-12-14; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Chronic Cough (CC)
Keywords: Pediatric; chronic cough; Etiologic Screening; Electronic Questionnaire
MeSH Terms: conditions — Chronic Cough | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Routine Care: Physician-Blinded to Questionnaire Results
  Interventions: Other: No intervention (observational study)
- Questionnaire-Assisted Care: Physician-Informed by Questionnaire Results
  Interventions: Other: No intervention (observational study)

INTERVENTIONS:
Other: No intervention (observational study) — No intervention (observational study)

SUMMARY:
Chronic cough is a common and burdensome condition in children, with complex and overlapping etiologies that often lead to delayed diagnosis, misdiagnosis, and inappropriate treatment. This prospective, controlled, observational study aims to develop and clinically validate a Wenjuanxing-based, parent-reported, multidimensional etiologic screening questionnaire for pediatric chronic cough. Children aged 3-18 years presenting with cough lasting ≥2 weeks will be enrolled in a tertiary pediatric respiratory clinic and allocated to either a routine-care group or a questionnaire-assisted group. All caregivers will complete the standardized electronic questionnaire, which generates an automated preliminary etiologic suggestion based on symptom patterns, triggers, and associated features. Diagnostic accuracy, treatment effectiveness, and symptom resolution will be evaluated through structured follow-up at two weeks. The primary outcome is the difference in diagnostic accuracy between physicians using routine assessment alone and those supported by the questionnaire. Secondary outcomes include treatment response and prevention of cough chronicity. This study seeks to provide evidence for a scalable, digital, and standardized screening tool to improve early etiologic identification and clinical decision-making in pediatric chronic cough.

DETAILED DESCRIPTION:
1. Development of a Wenjuanxing-based multidimensional etiologic screening questionnaire for pediatric chronic cough This study aims to develop and validate a structured, parent-reported, electronic questionnaire for multidimensional etiologic screening of chronic cough in children, based on current clinical practice guidelines and expert consensus. The questionnaire is designed and deployed on the Wenjuanxing platform and focuses on standardized, comprehensive, and reproducible symptom collection.

   The questionnaire includes multiple domains: cough duration and temporal pattern (daytime vs nocturnal cough), cough characteristics (dry vs wet), triggering factors (exercise, cold air, allergen exposure), associated respiratory and extra-respiratory symptoms (wheezing, nasal congestion, postnasal drip, throat clearing, gastroesophageal reflux symptoms), past medical history, family history, and environmental exposures. Logical branching and rule-based algorithms are embedded to automatically generate preliminary etiologic suggestions, including cough variant asthma (CVA), upper airway cough syndrome (UACS), protracted bacterial bronchitis (PBB), post-infectious cough (PIC), eosinophilic bronchitis (EB), and gastroesophageal reflux-related cough (GERC).

   The electronic format allows standardized data acquisition, real-time logic checking, automated output of etiologic suggestions, and efficient data export for subsequent clinical evaluation and statistical analysis.
2. Clinical validation of the questionnaire in routine outpatient practice This is a prospective, controlled, observational study conducted in the pediatric respiratory outpatient clinic of Shanghai Children's Medical Center. Children aged 3-18 years presenting with cough lasting ≥2 weeks and meeting the inclusion criteria will be consecutively enrolled after informed consent is obtained from their caregivers.

   All caregivers will complete the Wenjuanxing questionnaire. Participants will be assigned to one of two parallel groups according to the study protocol: a routine-care group, in which physicians perform diagnosis and treatment based on standard clinical assessment without access to questionnaire results; a questionnaire-assisted group, in which physicians review the questionnaire-generated etiologic suggestions before making diagnostic and therapeutic decisions.

   At the initial visit, physicians will record their clinical diagnosis and treatment plan. In the questionnaire-assisted group, physicians will additionally rate the perceived usefulness of the questionnaire and their level of confidence in the questionnaire's etiologic suggestions using standardized numeric scales.
3. Follow-up and outcome assessment All enrolled patients will be followed up approximately two weeks after the initial visit via telephone or online contact using a standardized operating procedure. Caregivers will be asked to report changes in cough symptoms, including degree of improvement, time to symptom relief, and overall treatment effectiveness. Caregivers will also rate the perceived consistency between the questionnaire-based etiologic suggestion and the physician's final diagnosis.

If symptom improvement is insufficient, further guidance and an additional follow-up may be conducted according to the study protocol. The primary outcome is the difference in diagnostic accuracy between the routine-care group and the questionnaire-assisted group, with follow-up response serving as post-hoc clinical validation. Secondary outcomes include treatment effectiveness, caregiver satisfaction, physician acceptance, and feasibility of implementing the questionnaire in real-world outpatient settings.

This study aims to establish a scalable, digital, and standardized screening approach for pediatric chronic cough, supporting early etiologic identification and improving clinical decision-making in routine practice.

ELIGIBILITY:
Inclusion CInclusion Criteria:

1. Children aged 3 to 18 years, any sex.
2. Presenting for medical care due to cough lasting ≥2 weeks.
3. No fever within the past 2 weeks.
4. Caregiver is willing to complete the Wenjuanxing questionnaire and agree to follow-up.

Exclusion Criteria:

1. Presence of congenital airway malformations, chronic lung disease, or severe immunodeficiency.
2. Recent participation in other interventional clinical research.
3. Unable to complete follow-up as required.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children aged 3 to 18 years presenting to the pediatric respiratory outpatient clinic of Shanghai Children's Medical Center with cough lasting at least 2 weeks will be eligible for enrollment. The study population consists of symptomatic pediatric patients without fever in the preceding two weeks, whose caregivers are willing to complete an electronic questionnaire and participate in follow-up assessments. Participants will receive routine clinical evaluation and management according to standard practice, with or without access to questionnaire-generated etiologic suggestions, depending on study group assignment.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Accuracy of Initial Etiologic Assessment for Pediatric Chronic Cough | Approximately 2 weeks after the initial outpatient visit
  Diagnostic accuracy is defined as the concordance between the initial etiologic diagnosis made at the first outpatient visit and the post hoc clinical validation based on symptom response during follow-up. Caregivers will be contacted approximately two weeks after the initial visit and asked to report changes in cough symptoms using a standardized follow-up protocol. An initial diagnosis will be considered correct if the prescribed treatment results in marked improvement or resolution of cough symptoms, as assessed by caregiver-reported symptom improvement and overall treatment effectiveness. The diagnostic accuracy will be compared between the routine-care group and the questionnaire-assisted group.

CONTACTS AND LOCATIONS:
Overall Officials: Yong Yin, PhD, Principal Investigator — Shanghai Children's Medical Center
Locations (1):
- Shanghai Children's Medical Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided